CLINICAL TRIAL: NCT00618488
Title: Clinical Efficacy of Yogurt Containing Bifidobacterium Lactis (BB12) in Subjects With Functional Gastrointestinal Symptoms
Brief Title: Efficacy of Yogurt Containing BB12 in Subjects With GI Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina (Other)
Collaborators: General Mills (Industry)
Responsible Party: Yehuda Ringel M.D./Principal Investigator, Center for Digestive Diseases and Nutrition
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-0922
Record Dates: First submitted 2008-02-07; First posted 2008-02-20 (Estimated); Last update posted 2008-02-20 (Estimated); Status verified 2008-02

CONDITIONS: Pain
Keywords: Probiotics; BB12; Gastrointestinal Symptoms
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Bifidobacterium lactis
  Interventions: Dietary Supplement: Probiotic BB12 - Bifidobacterium lactis
- 2 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic BB12 - Bifidobacterium lactis — Bifidobacterium lactis (3.1 oz yogurt) administered once a day for 6 weeks
  Arms: 1
Dietary Supplement: Placebo — Placebo administered once a day for 6 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to determine if probiotics bacteria, specifically bifidobacterium lactis (BB12) improve gastrointestinal symptoms in subjects with functional gastrointestinal symptoms (i.e., non-patients IBS/functional bowel disorders).

DETAILED DESCRIPTION:
The apparent success of the use of probiotics in several gut disorders (e.g., IBD and rotavirus diarrhea) together with the greater understanding of the role of inflammation and intestinal microflora in the pathophysiology of functional bowel disorders has led to increased interest in use of probiotics in patients with these symptoms. The data on the use of probiotic in certain functional GI disorders (e.g., IBS, bloating, diarrhea) is limited but several reported studies show encouraging results and suggest some symptomatic response and parallel improvement in quality of life. Functional Bowel Disorders (FBD) - According to the Rome II criteria FBD refer to symptoms attributed to the mid or lower GI tract. FBD include several clinical subgroups including irritable bowel syndrome (IBS), functional diarrhea, functional constipation, functional abdominal bloating, and an unspecified group. This study will examine 'Non-Patients IBS,' these are people who have functional gastrointestinal (GI) symptoms but do not sought out medical care for their GI symptoms and therefore they are referred to as 'Non-patients'. This study will investigate the overall effect of probiotic bacteria (BB12) on GI symptoms in non-patients subjects with functional bowel symptoms (FBS).

ELIGIBILITY:
Inclusion Criteria:

* The subject is 18 - 70 y/o.
* The subject has any functional GI symptoms that are related to IBS, functional diarrhea, functional constipation, or functional bloating according to the Rome II criteria for functional GI disorders. The subject has the above symptoms for at least two weeks (i.e., active symptoms on enrollment). The subject has not been seen by a medical care provider for these symptoms in the 10 months and is not taking prescribed medications for these symptoms. Over the counter (OTC) medications are allowed as long as the subject is still symptomatic despite current OTC therapy.
* For diarrhea we will use the definition of a mean of >2 bowel movements per day, or a mean score of > 4 on the Bristol Stool Form Scale per week.
* For constipation we will use the definition of a mean of <3 bowel movements per week or a need for significant straining for a bowel movement.
* The subject's symptoms are mild to moderate in severity. Symptoms severity will be assessed at baseline and at the end of the 2-weeks screening period to determine eligibility prior randomization. Severity of bowel symptoms will be determined using the Francis Whorwell IBS severity scale: Mild <175, Moderate 175-300, Severe >300
* Subject must have had a normal colonoscopy within the last 3 years if age >50y/o.
* Subjects' initial evaluation at screening visit including medical history, physical examination, and laboratory tests are unrevealing i.e., do not show abnormalities that require further investigation.

Exclusion Criteria:

* The subject saw a physician for your functional bowel symptoms in the last 10 months
* The subject has taken prescribed medications for your functional bowel symptoms
* The subject has inflammation or structural abnormality of the digestive tract [e.g. inflammatory bowel disease (IBD), duodenal ulcer (DU) or gastric ulcer (GU), obstruction, or symptomatic cholelithiasis].
* The subject has severe FBD symptoms at baseline.
* The subject carries a medical diagnosis of FBD and has seen a medical care provider and take prescribed medications for their GI symptoms. Patients who did not see a medical care provider for these symptoms for more than 10 months and are not taking prescribed medications for their GI symptoms are eligible.
* The subject has a serious, unstable medical condition.
* The subject has insulin-dependent Diabetes Mellitus.
* The subject had a major psychiatric diagnosis or a suicide attempt within the last two years.
* The subject has a history of alcohol or substance abuse within two years.
* The subject has abnormal laboratory results (including ALT or AST > than 2.5 times normal, serum creatinine >2.0mg/dl, untreated abnormal TSH value)
* The subject has been treated for a malignancy within the last 5 years (except BCC or SCC skin cancer).
* The subject has been diagnosed with lactase deficiency and this can explain their symptoms (i.e., symptoms resolved or reduced significantly with lactose-free diet.)
* The subject has participated in a drug study within the last 21 days.
* The subject received antibiotic treatment or intentionally consumes probiotic products during the last 6 weeks. (If the subject was on antibiotic or probiotics treatment, a washout period of 6 weeks is required).
* The subject had previous significant gastric or intestinal surgery.
* Patient is pregnant or lactating due to possible effects of hormonal changes during pregnancy on GI functions and/or functional GI symptoms.
* The subject is predisposed to infection (i.e. their immune system is compromised, they have rheumatic heart disease, an artificial valve, history of bacterial endocarditis, or an active bacterial disease).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The global relief of functional GI symptoms as assessed by Global Symptom Assessment (GSA) of relief of functional GI symptoms. | March 2008

SECONDARY OUTCOMES:
The satisfaction with treatment as assessed by Satisfaction Survey. | March 2008

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ringel, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States